CLINICAL TRIAL: NCT04330131
Title: TMW Center for Early Learning + Public Health Community-Wide Demonstration Project
Brief Title: TMW Community-Wide Demonstration Project
Acronym: TMW-CWDP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges due to covid prevented implementation of this behavioral study in a hospital setting
Sponsor: University of Chicago (Other)
Collaborators: Childrens Services Council (Unknown); St. Mary's Medical Center (Other); Soma Medical Center (Unknown); HomeSafe (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-1588
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Language Development

STUDY DESIGN:
Intervention Model Description: Treatment group participants will consist of all the families who enroll in the TMW interventions in the hospitals and clinics of the treated community (the target zip codes for intervention delivery). The comparison group will consist of families enrolled from hospitals and pediatric clinics with similar characteristics to the treatment group sites.Then within this comparison group, the researchers will define a sample of comparison families who have similar individual characteristics as the treated families.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated families (Experimental): The treated families will complete up to 3 interventions: 3Ts - Newborn, 3Ts - Well Baby, and 3Ts - Let's Talk! The ideal progression is that treated families will complete all three interventions. Before completing their first intervention, participants will complete set of baseline surveys measuring their knowledge and beliefs about child development. They will repeat these measures when their child is 6 months, 9 months, 1-, 2-, and 3-years old.
  Interventions: Behavioral: 3Ts - Newborn; Behavioral: 3Ts - Well Baby; Behavioral: 3Ts - Let's Talk!
- Comparison Families (No Intervention): Comparison families will not receive any of the 3Ts interventions but will complete the same surveys as the treatment group at study enrollment and again when their child is 6 months, 9 months, 1-, 2-, and 3-years old.

INTERVENTIONS:
Behavioral: 3Ts - Newborn — A video shared with parents/caregivers during a universal screening in hospital mother-baby units. This intervention shares the importance of early talk and interaction with a child to support their early brain development as well as strategies for parents to do so.
  Arms: Treated families
Behavioral: 3Ts - Well Baby — Four videos shared during well child immunization visits at 1-, 2-, 4-, and 6-months in pediatrician offices. This intervention shares the importance of early talk and interaction with a child to support their early brain development as well as strategies for parents to do so.
  Arms: Treated families
Behavioral: 3Ts - Let's Talk! — A series of eight group classes involving education, feedback, and goal setting for parents/caregivers of children age one through three, delivered in a community-based organization. This intervention shares the importance of early talk and interaction with a child to support their early brain development as well as strategies for parents to do so.
  Arms: Treated families

SUMMARY:
The TMW Center is launching a community-wide demonstration project in partnership with the Children's Services Council of Palm Beach County, Florida, in which the TMW interventions will be delivered at scale through partners who work with families across health, education, and social service systems. The goal of this partnership is to reach 60% of all families with children age birth through three with at least one TMW intervention over the five-year partnership, with a significant percentage of families receiving more than one intervention. The TMW Center will evaluate the efficacy of the multiple intervention approach in impacting parent knowledge, beliefs, and behavior and child developmental outcomes, and develop an implementation model that can be used in other communities.

DETAILED DESCRIPTION:
The treatment community will consist of all participants enrolled in one or more of the 3Ts Interventions (3Ts-Newborn, 3Ts-Well Baby, 3Ts-Let's Talk!) The 3Ts interventions, the educational curricula designed by the TMW Center) were named for the three easy to use strategies that are shared with parents to support their child's development: Tune In, Talk More, and Take Turns.

To compare outcomes and evaluate effectiveness of the interventions, a comparison community will be selected beginning in 2021. To define the sample of comparison families, the TMW Center and CSC will work to find a comparison hospital with similar socioeconomic characteristics and child developmental outcomes as the treated community. Then within this comparison group, the researchers will define a sample of comparison families who have similar individual characteristics as the treated families (based on data shared by CSC and baseline data the researchers will collect). They will complete the same surveys as the treatment community but will not be offered the interventions.

The following describes the ideal progression through the full intervention and study timeline. However, participants are able to join during any intervention time point (e.g. 3Ts-Newborn, or the third 3Ts-Well Baby video time point, etc), even if they have not completed previous study measures. Whenever a participant engages 3Ts interventions for the first time, they will complete the eConsent module prior to receiving any intervention content. They will complete only the surveys applicable to the time point of their enrollment and beyond, according to the study timeline. Similarly, if they choose to skip certain interventions or survey time points, they will still be able to complete the later time points. The researchers will not ask participants to complete any missed intervention or survey time points or require them to complete any skipped interventions or surveys. Participants selected in the comparison group will complete only the activities here labeled 'Data Collection.'

Data collection: Baseline These measures will be collected at the parent's first interaction with the TMW study, regardless of intervention time point. Following the eConsent, participants will be asked to provide contact information and basic demographic information (parent name, parent DOB, child DOB). Then participants will be asked to fill out one survey, the Survey of Parental Expectations and Knowledge about Language Learning (SPEAK) that assess their knowledge and beliefs of child language and cognitive development. The version of the SPEAK to be used will depend on the child's age and at which intervention they are completing the baseline measures. If the participant's baseline is at the 3Ts-Newborn Intervention, the parent will complete SPEAK-20. If done at the start of the 3Ts-Well Baby Intervention, participants will complete the Baby SPEAK-10. eConsent and surveys will be collected digitally through the secure online platform.

Intervention 1: 3Ts-Newborn This intervention is completed with parents of newborns in the postpartum mother-baby unit in the hospital. Participants will complete the 3Ts-Newborn educational intervention as part of Florida's Universal Infant Screen. After completing the eConsent module and filling out the demographics survey, parents will complete the SPEAK-20 survey using the tablet. After this, they will watch the 12 minute education intervention video, also on the tablet. Finally, parents will complete the Baby SPEAK-10 survey using the tablet.

Intervention 2: 3Ts-Well Baby The 3Ts-Well Baby Intervention will take place in pediatricians' offices during regularly scheduled well child immunization appointments. All parents with a child under 7 months of age who are receiving care at participating locations will be offered the opportunity to complete a video intervention module at their child's appointment from the ages of 1 to 6 months. This intervention will take place entirely on a tablet. If a participant did not complete the 3Ts-Newborn intervention, they will complete the eConsent module, demographics survey, and the Baby SPEAK-10 survey prior to viewing the first educational module. Parents who return for multiple well-child appointments while the child is 6 months or younger may complete up to a total of 4 educational video modules, one per visit.

Data collection: 6 months At age six months participants will be asked to fill out the Baby SPEAK-10 and PACOTIS surveys, either onsite at their pediatric visit via the tablet provided by CSC partners or at home by logging into the TMW Tech Platform. The PACOTIS is a self-report measure of the respondent's perceived impact on their child's development. Participants in the treatment community will have access to the surveys upon completion of the fourth 3Ts-Well Baby Intervention Video, while participants in the comparison group will receive a notification from the TMW Tech Platform that it is time to complete the surveys. These surveys will take approximately 10 minutes to complete.

Data collection: 9 months At age nine months, all participants will be asked to fill out two surveys, the Baby SPEAK-10 and the PACOTIS. All participants will receive a notification from the TMW Tech Platform that it is time to complete the surveys. These surveys, which are completed through the TMW Tech Platform, will take approximately 10 minutes to complete.

Intervention 3: 3Ts-Let's Talk! Beginning in 2021, the 3Ts-Let's Talk! intervention will be offered to parents who engage in CSC community-based programming at any time their child is 0-3 years old. Participants need not have completed previous interventions to be part of this intervention, and if this is their first interaction with TMW, will complete the eConsent module, demographics survey, and SPEAK-10. 3Ts-Let's Talk! will take place at partnering community organizations and participants will review educational modules with other parents in a group setting.

Data collection: 12 months Two weeks before the child turns 12 months, participants will be receive a notification from the TMW Tech Platform that it is time to complete their next surveys. They will be asked to complete the Baby SPEAK - 10 and the StimQ-Reading Subscale. The StimQ is a parent report measuring parental verbal responsivity and involvement in their child's development.

Two weeks after the child turns 12 months, participants will receive another notification from the TMW Tech Platform asking them to complete a second set of surveys, consisting of the MacArthur-Bates Communicative Development Inventories: Short Form Level 1 (MCDI I-SF) and the PACOTIS. The MCDI I-SF is a parent report assessing children's vocabulary comprehension and production, appropriate for children 8-18 months. These surveys, which are again completed through the TMW Tech Platform, will take approximately 10 minutes to complete.

Data collection: 24 months Two weeks before the child turns 24 months, participants will receive a notification from the TMW Tech Platform that it is time to complete their next surveys. They will be asked to complete the SPEAK-10 and the StimQ-Reading Subscale. These surveys, which are completed through the TMW Tech Platform, will take approximately 10 minutes to complete.

Two weeks after the child turns 24 months, participants will receive another notification from the TMW Tech Platform asking them to complete a second set of surveys, consisting of the MacArthur-Bates Communicative Development Inventories: Short Form Level 2 (MCDI II-SF) and the PACOTIS. The MCDI II-SF is an extension of the MCDI-I-SF and is appropriate for ages 16-30 months. These surveys, which are completed through the TMW Tech Platform, will take approximately 10 minutes to complete.

Data collection: 36 months Two weeks before the child turns 36 months, participants will receive a notification from the TMW Tech Platform that it is time to complete their next surveys. They will be asked to complete the SPEAK-10 and the StimQ-Reading Subscale. These surveys, which are completed through the TMW Tech Platform, will take approximately 10 minutes to complete.

Two weeks after the child turns 36 months, parents will receive another notification from the TMW Tech Platform asking them to complete a second set of surveys, consisting of the MacArthur-Bates Communicative Development Inventories: Short Form Level 2 (MCDI II-SF) and the PACOTIS. Spanish speaking participants will not complete the MCDI II-SF at 36 months, because the Spanish version does not go beyond 30 months, while an extension to 37 months has recently been developed in in English. These surveys, which are completed through the TMW Tech Platform, will take approximately 10 minutes to complete.

Between study activities, participants will receive text messages to the phone number they provide. These text messages will be content nudges to remind participants of ways they can use the strategies learned throughout the interventions in their day to day life. For example, "remember to use the 3Ts to build baby's brain while driving to school!"

Participants will also have online access to additional educational videos and resources. These resources are optional and parents can view as many or as few as they wish throughout the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be able to understand English or Spanish
* Must be the parent/caregiver of a child in the target range of the intervention (at birth for the 3Ts-Newborn, 0-6 months for 3Ts-Well Baby and 0-3 years for 3Ts-Let's Talk!). For this study, the parent is defined as person with custody of the child.

Exclusion Criteria:

* Parents under the age of 18 who are not emancipated minors
* Parents who do not have legal custody of their child
* Parents who do not speak enough English or Spanish to receive their educational information in that language.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Survey of Parental Expectations and Knowledge (SPEAK) | Up to 3-years of age
  Measures parental knowledge and expectations of how their children learn language at different ages. Some items about beliefs of appropriate age of exposure are rated on a 6-point scale ranging from: 1 "As an infant (0 to 6 moths)" to 6 "In elementary school (6 years and up)" Other items are rated on a 4-point Likert scale ranging from 1 (definitely true), 2 (probably true), 3 (probably not true) to 4 (definitely not true). Scores range from 0 to 71, and scoring of each item is based a criterion scale, with 0 points given to the most incorrect response and 1 additional point given to each progressively more correct response. A higher score correlates to a better outcome and indicates a higher parental knowledge.
Parental Cognition and Conduct Toward the Infant Scale (PACOTIS) | Up to 3-years of age
  A self-report measure of the respondent's perceived impact on their child's development. Scores for each of the 5 items range from 0 ('Not at all what I think') to 10 ('Exactly what I think'). A lower score indicates a better outcome
MacArthur-Bates Communicative Development Inventories-Short Form (MCDI-SF) | Up to 3-years of age
  Parent report measure of words that their child understands and says. For a list of words, a parent marks whether a child 'understands', 'understands and says' or 'neither understands nor says.' Each column is tallied and higher counts in the 'understands and says' column indicate better outcomes
StimQ - Reading Subscale | Up to 3-years of age
  A questionnaire that is designed to explore the different kinds of activities that primary caregivers engage in with their infant child, preschool child, or toddler and their role in promoting cognitive stimulation for the child. Items 1-4 are scored on a scale of 0-4 based on how often a parent engages in certain behaviors. Items 5-10 are scored as a Yes (1 point) or No (0 points). A higher score indicates a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dana Suskind, M.D., Principal Investigator — University of Chicago
Locations (4):
- United States (4):
  - Soma Medical Center, PA #3-Forest Hill, West Palm Beach, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Soma Medical Center, PA#4 Military, West Palm Beach, Florida
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suskind DL, Leffel KR, Graf E, Hernandez MW, Gunderson EA, Sapolich SG, Suskind E, Leininger L, Goldin-Meadow S, Levine SC. A parent-directed language intervention for children of low socioeconomic status: a randomized controlled pilot study. J Child Lang. 2016 Mar;43(2):366-406. doi: 10.1017/S0305000915000033. Epub 2015 Jun 4. PMID 26041013
- See also: The homepage for the TMW Center for Early Learning and Public Health — https://tmwcenter.uchicago.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04330131/Prot_SAP_000.pdf